CLINICAL TRIAL: NCT06233136
Title: Effect of Leg Pedalling Exercise From Inclined Position on Functional Ability and Trunk Control in Children With Diplegic Cerebral Palsy
Brief Title: Effect of Leg Pedalling Exercise From Inclined Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Bahgat mahmoud Hasan, Scientific researcher, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004085
Record Dates: First submitted 2023-07-24; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Palsy Spastic Diplegia
Keywords: Leg Pedalling
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leg Pedalling exercise and designed physical therapy program (Experimental): Each child in the experimental group will be positioned in semi-reclined position with 45 degree trunk flexion during the application of cycling Sessions will be 30 minutes per session, three times per week, for two successive months The designed physical therapy program It will be applied for all participated children in both groups. It includes;
  1. Flexibility exercises
  2. Static and dynamic balance exercises
  3. Functional training Sessions will be 45 minutes per session, three times per week, for two successive month
  Interventions: Device: Leg pedalling exercise; Other: The designed physical therapy program
- Designed physical therapy program (Active Comparator): The designed physical therapy program It will be applied for all participated children in both groups. It includes;
  1. Flexibility exercises
  2. Static and dynamic balance exercises
  3. Functional training Sessions will be 45 minutes per session, three times per week, for two successive month
  Interventions: Other: The designed physical therapy program

INTERVENTIONS:
Device: Leg pedalling exercise — Each child in the experimental group will be positioned in inclined position and will cycle through the range of motion under the supervision of the researcher
  Other Names: Leg ergometer
  Arms: Leg Pedalling exercise and designed physical therapy program
Other: The designed physical therapy program — It applied for all participated children in both groups. It includes;
  1. Flexibility exercises
  2. Static and dynamic balance
  3. Functional training exercises
  Other Names: Traditional physical therapy program

SUMMARY:
Statement of the problem:- Does the lower limb pedalling exercise from inclined position improve functional ability and trunk control in children with diplegic cerebral palsy? Null Hypothesis:- There will be no effect of lower limb pedalling exercise from inclined position on functional ability and trunk control in children with diplegic cerebral palsy

DETAILED DESCRIPTION:
Subjects A convenient sample of children diagnosed as spastic diplegic cerebral palsy (CP) from both sexes will be recruited based on a pilot study according to the inclusion and exclusion criteria. They will be selected from the out-patient private clinics in Giza and Tenth of Ramadan City.

Study design:

Randomized controlled clinical trial. Children will receive intervention type randomly, 15 child received the designed physical therapy program and the pedaling exercise from inclined position and the other 15 child receieved the designed physical therapy program only. Children will be assessed by measuring functional ability with Gross Motor Functional measures and trunk control with trunk control measurement scale

ELIGIBILITY:
Inclusion Criteria:

.Age ranges from 6-9 years. .Grade 1, 1+ of the Modified Ashworth Scale.

.Level II, III according to Gross MotorFunctional Classification System (GMFCS).

.Able to pedal independently on a static bicycle.

.Ability to follow command.

Exclusion Criteria:

.Significant visual or auditory impairments.

.Structural or fixed deformities of lower extremities.

.Perception disorders.

.Botox injection in the lower extremity in the past 6 months.

.Lower extremity surgery within the past 6 months.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
The gross motor function scale | 2 months for each participant
  Assessment of change of functional ability carried out by using gross motor function measures
Assessment of trunk control | 2 months for each participant
  Assessment of change of trunk control carried out by using trunk control measurement scale

CONTACTS AND LOCATIONS:
Overall Officials: NANEES E Mohamed, Phd, Study Director — Professor
Locations (1):
- Faculty of physical therapy cairo University, Dokki, Giza Governorate, Egypt